CLINICAL TRIAL: NCT05578443
Title: Efficacy, Safety and Response Predictors of Astragalus Membranaceus on the Improvement of Cognitive Function in Mild-to-Moderate Alzheimer's Disease: a Randomized Controlled Trial Protocol
Brief Title: Efficacy, Safety and Response Predictors of Astragalus Membranaceus on the Improvement of Cognitive Function in Mild-to-Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AD-AS
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10g Astragalus membranaceus (Experimental)
  Interventions: Drug: 10g Astragalus; Behavioral: Routine treatment
- Routine treatment (Experimental)
  Interventions: Behavioral: Routine treatment
- 20g Astragalus membranaceus (Experimental)
  Interventions: Behavioral: Routine treatment; Drug: 20g Astragalus

INTERVENTIONS:
Drug: 10g Astragalus — Astragalus tablets 10g, warm water to drink, once a day, take for 1 year, during which routine treatment should also be carried out.
  Arms: 10g Astragalus membranaceus
Behavioral: Routine treatment — Limit water and sodium intake. Raise the head of the bed. Standardized amount of exercise. Low temperature diet and small meals. Avoid alcohol, coffee and dehydration. The treatment lasted for 3 months.
Drug: 20g Astragalus — Astragalus tablets 20g, warm water to drink, once a day, take for 1 year, during which routine treatment should also be carried out.
  Arms: 20g Astragalus membranaceus

SUMMARY:
Alzheimer's disease (AD), the most common cause of dementia, is characterized by cognitive impairment, mental and behavioural abnormalities, and social dysfunction. Current treatments can only delay the progression of AD, not cure it completely. In vitro studies have shown that Astragalus has toxic effects such as anti-hypoxia injury of nerve cells, anti-free radical damage, anti-excitatory amino acids, etc. It can be used to expand cerebral vessels, increase cerebral blood flow, improve cerebral microcirculation, protect brain cells, and repair damaged brain cells. However, the clinical effects of add-on Astragalus in improving cognition in these patients remain unclear. Therefore, this pragmatic clinical trial aims to determine the efficacy and safety of add-on Astragalus in improving cognition in patients with AD

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be as follows:

1. Male or female aged ≥50 years and ≤85 years
2. Memory loss for at least 6 months, with a progressive worsening trend Patients with mild or moderate disease degree, that is, the total score of MMSE: 14 points < total score of MMSE <24 points, 0.5≤CDR≤2 points, and the total score of HAMD (24-item version) ≤20 points
3. Brain magnetic resonance imaging shows the degree of hippocampal atrophy is greater than or equal to grade 1
4. The modified Hachinski Ischemia Scale (m-HIS) score was < 4 points
5. The criteria described by the diagnostic and statistical manual of mental disorder-V for the diagnosis of dementia comply with the National Institute on Aging - Alzheimer's Association "Very likely AD" (National Institute of Aging-Alzheimer's Association, 2011).
6. There are no obvious positive signs in nervous system examination;
7. The subjects have the ability of reading, writing and communication, have a stable caregiver, accompany to attend the visit.
8. The basic treatment of AD before enrollment remained unchanged, and if long-term users needed to use it steadily for more than 4 weeks before randomization,the dose was kept as stable as possible during the study. Such drugs include: cholinesterase inhibitors.

Exclusion Criteria:

The exclusion criteria will be as follows:

1. MRI showed significant focal lesions, including one of the following: a. There were more than 2 infarcts with a diameter greater than 2cm; b. Infarcts in key areas such as the thalamus, hippocampus, entorhinal cortex, parorhinal cortex, angular gyrus, cortex, and other subcortical gray matter nuclei; c. White matter lesion Fazekas Scale ≥3
2. Patients who have taken other Chinese medicine preparations in the past three months
3. Allergy or contraindication of astragalus
4. There are other neurological diseases that can cause brain dysfunction or cognitive impairment; Mental and neurological retardation is present; Presence of malignant tumor
5. The modified Hachinski Ischemia Scale (m-HIS) score was ≥ 4 points. Patients who refuse or have MRI or EEG contraindications (pacemakers, coronary and peripheral arterial stents, Metal implants, claustrophobia, or severe visual or hearing impairment), refusing to draw blood
6. Pregnant or lactating patients;
7. Patients who have participated in other clinical studies within the past 3 months

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy outcome measure will be the absolute change in the Alzheimer's Disease Assessment Scale-Cognitive Subscale, Chinese version score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale, Chinese version scale scores range from 0 to 75, with higher scores indicating better.

SECONDARY OUTCOMES:
The absolute scores change in the Rey-Osterrieth Complex Figure Test [ROCF] recall score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline
  The ROCF scale scores range from 0 to 36, with higher scores indicating better.
The absolute scores change in the ROCF-copy score between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  The ROCF copy scale scores range from 0 to 36, with higher scores indicating better.
The absolute scores change in the Clock-Drawing Test score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline
  The Clock-Drawing Test scale scores range from 0 to 5, with higher scores indicating better.
The absolute scores change in the Trail Making Test-A score between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  The Trail Making Test-A scores range from 0 to 25, with higher scores indicating better.
The absolute scores change in the Digit Span Forward score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  TheDigit Span Forward score scores range from 0 to 10, with higher scores indicating better.
The absolute scores change in the Trail Making Test-B score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Trail Making Test-B scores range from 0 to 25, with higher scores indicating better.
The absolute scores change in the Digit Span Backward score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Digit Span Forward score scores range from 0 to 9, with higher scores indicating better.
The absolute scores change in the Verbal Fluency Test score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Verbal Fluency Test score scores range from 0 to 14, with higher scores indicating better.
The absolute scores change in the Hamilton Anxiety Scale score between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  The Hamilton Anxiety Scale score scores range from 0 to 56, with higher scores indicating worse.
The absolute scores change in the Hamilton Depression Scale score between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  The Hamilton Anxiety Scale score scores range from 0 to 96, with higher scores indicating worse.
The absolute change in the blood pressure between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  To observe the changes of orthostatic blood pressure in patients
The absolute change in the level of plasma β-amyloid40 (ng/ml) between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Amyloid is one of the main biomarkers of dementia
The absolute change in the level of plasma β-amyloid42 (ng/ml) between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  Amyloid is one of the main biomarkers of dementia
The absolute change in the level of plasma glial fibrillary acidic protein (ng/ml) between baseline and week 48 | Participants will be followed up for 48 weeks after baseline
  Glial fibrillary acidic protein is one of the main biomarkers of dementia
The absolute change in the level of plasma neurofilament light chain (ng/ml) between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Neurofilament light chain is one of the main biomarkers of dementia
The absolute change in the level of plasma hyper-phosphorylated tau-181 (ng/ml) between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  Neurofilament light chain is one of the main biomarkers of dementia
The absolute change in the P300 between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  P300 is the main indicator of EEG, and its normal value range is between 320 and 420
The absolute change in the VP300 between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  VP300 is the main indicator of EEG, and its normal value range is between 320 and 420.
The absolute change in the MMN between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  MMN is the main indicator of EEG, and its normal value range is between 100 and 210.
The absolute change in the neurite density index between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  Neurite density index is the main indicator of neurite-oriented diffusion and density imaging (NODDI) .
The absolute change in the orientation dispersion index between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  Orientation dispersion index is the main indicator of neurite-oriented diffusion and density imaging (NODDI) .
The absolute change in the isotropic volume fraction between baseline and week 48 | Participants will be followed up for 48 weeks after baseline.
  Isotropic volume fraction is the main indicator of neurite-oriented diffusion and density imaging (NODDI) .
The absolute change in surface area between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Surface area is the main indicator of voxel-based morphometry.
The absolute change in thickness, between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Thickness, is the main indicator of voxel-based morphometry.
The absolute change in volume, between baseline and week 48. | Participants will be followed up for 48 weeks after baseline.
  Volume, is the main indicator of voxel-based morphometry.

OTHER OUTCOMES:
Whether the participants' vital signs were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Whether the participants' Electrocardiograms were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Whether the participants' Liver function were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Whether the participants' kidney function were normal. | Participants will be followed up for 48 weeks after baseline.
  Safety outcome
Severity of adverse events | Participants will be followed up for 48 weeks after baseline.
  Safety outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No